CLINICAL TRIAL: NCT06740396
Title: Assessing the Prevalence and Severity of Depression Among Coronary Artery Diseases Patients in Baghdad Using the PHQ-9: A Cross-Sectional Study
Brief Title: Prevalence and Severity of Depression in Coronary Artery Disease Patients
Acronym: PAD-CAD
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241214; 016 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Depression - Major Depressive Disorder
Keywords: PHQ-9

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This observational study aims to estimate the prevalence and severity of depression among patients with coronary artery disease (CAD) in Baghdad, Iraq, using the self-administered PHQ-9 questionnaire. The study seeks to answer the following questions:

What is the prevalence of depression among CAD patients? How is the severity of depression distributed within this group? Are specific demographic, clinical, or environmental factors associated with higher levels of depression?

Participants will:

Complete the PHQ-9 to assess the severity of depressive symptoms at a specific point in time.

Provide demographic and clinical information, including age, gender, socioeconomic status, comorbidities, and CAD-related factors such as type of intervention and duration of illness, to explore potential correlations with depression.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) remains one of the leading causes of morbidity and mortality worldwide, with multiple risk factors influencing its onset and progression. Among the psychosocial factors associated with CAD, depression plays a particularly prominent role. Research indicates that while 17% to 27% of patients with CAD have major depression, a significantly larger percentage experience subsyndromal depressive symptoms. This highlights a widespread issue where depressive symptoms, even if not clinically classified as major depression, still contribute to poorer health outcomes in CAD patients. Major depression is not only prevalent among CAD patients but is also linked to an increased risk for developing CAD and higher mortality from the disease. However, the exact mechanisms through which depression impacts cardiovascular health remain unclear.

Coronary heart disease (CHD), a major manifestation of CAD, typically results from the rupture or erosion of an atherosclerotic plaque in the epicardial coronary arteries. Over 60 risk factors and markers have been associated with the initiation and progression of these plaques. When a plaque ruptures, it can stimulate acute thrombosis within the artery, leading to an acute coronary syndrome (ACS), which may present as a myocardial infarction (MI), unstable angina, or even sudden cardiac death. These risk factors can be broadly categorized into three groups: lifestyle, biological, and psychosocial. Depression, as a psychosocial risk factor, not only increases the likelihood of developing CAD but also contributes to worse outcomes in patients who already have the disease.

The impact of depression extends beyond its role in the progression of CAD; it significantly affects the quality of life (QOL) of patients with coronary disease. While treating depression may not necessarily reduce depression's role as a direct risk factor for CAD, improving the quality of life should be considered a primary goal of treatment. Defining and measuring QOL remains a challenge, but recent studies have shown a clear relationship between QOL, depression, and mortality risk in CAD patients. This underscores the importance of addressing both the psychological and physical health of CAD patients in clinical care.

Moreover, the PHQ-9 (Patient Health Questionnaire-9) is a widely used, self-administered tool designed to assess the severity of depression in individuals. Comprising nine simple, straightforward questions, the PHQ-9 evaluates the frequency of common depressive symptoms over the past two weeks, such as feelings of sadness, loss of interest, sleep disturbances, and fatigue. Each response is scored on a scale from 0 to 3, and the total score helps determine the severity of depression, ranging from minimal to severe. Originally developed as a screening tool, the PHQ-9 is now a key instrument in both clinical practice and research for diagnosing major depressive disorder (MDD), monitoring treatment progress, and identifying individuals at risk for worsening symptoms. A meta-analysis conducted in 2015, which included 36 studies with over 21,000 participants, evaluated the sensitivity and specificity of various cut-off scores ranging from 7 to 15. The analysis found that the standard cut-off of 10 had a pooled sensitivity of 0.78 and specificity of 0.87, suggesting it is a reasonably effective screening tool. However, the study also noted significant limitations, such as incomplete reporting on cut-off scores other than 10, which led to misleading results indicating that sensitivity increased with higher cut-off scores, possibly due to selective reporting in some studies.

Despite the well-established connection between depression and CAD in many parts of the world, there is a notable gap in research on this topic within Iraq. This study aims to assess the prevalence and severity of depression among CAD patients in Baghdad using the Patient Health Questionnaire-9 (PHQ-9), a widely recognized tool for diagnosing depression. By exploring the burden of depression in this patient population, this research will provide important insights into the mental health needs of CAD patients in Iraq and contribute to improving both cardiovascular outcomes and quality of life in this underserved region.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with coronary artery disease (confirmed through clinical, imaging, or procedural evidence).
* Receiving care at designated hospitals in Baghdad.
* Able to understand and complete the PHQ-9 questionnaire independently or with minimal assistance.
* Consents to participate in the study.

Exclusion Criteria:

* Patients with a history of severe psychiatric disorders unrelated to depression (e.g., schizophrenia, bipolar disorder).
* Patients with cognitive impairments or neurological conditions affecting their ability to complete the questionnaire.
* Those currently hospitalized for acute cardiac events (e.g., myocardial infarction) requiring intensive care.
* Individuals unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients diagnosed with coronary artery disease (CAD) who are receiving outpatient or inpatient care in selected hospitals in Baghdad, Iraq. Participants will represent a diverse population in terms of age, gender, socioeconomic status, and comorbid conditions. The study aims to capture the prevalence and severity of depression within this group, considering the physical and psychological burden associated with CAD. Efforts will be made to recruit a representative sample to ensure that findings are generalizable to the broader population of CAD patients in Baghdad.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Depression | Data collection will occur over a 3-month period, with each participant completing the assessment at a single point during this time frame.
  Proportion of coronary artery disease patients in Baghdad who exhibit depressive symptoms.
Severity of Depression | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  The severity of depression in this study will be determined based on the scores obtained from the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 categorizes depression severity as follows: Minimal depression: Scores 0-4, indicating little to no symptoms. Mild depression: Scores 5-9, suggesting occasional symptoms that may not significantly affect daily functioning. Moderate depression: Scores 10-14, indicating more frequent symptoms that can interfere with daily life. Moderately severe depression: Scores 15-19, showing pronounced symptoms that significantly impact daily activities. Severe depression: Scores 20-27, with symptoms that are debilitating.
Patient Health Questionnaire-9 (PHQ-9) | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  The total score can range from 0 to 27. Higher scores indicate greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Aws Al-Rubaye Lecturer, Internal Medicine, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akosile W, Tiyatiye B, Colquhoun D, Young R. Management of depression in patients with coronary artery disease: A systematic review. Asian J Psychiatr. 2023 May;83:103534. doi: 10.1016/j.ajp.2023.103534. Epub 2023 Feb 28. PMID 36871435
- [Background] Bremner JD, Campanella C, Khan Z, Fani N, Kasher N, Evans S, Reiff C, Mishra S, Ladd S, Nye JA, Raggi P, Vaccarino V. Brain mechanisms of stress and depression in coronary artery disease. J Psychiatr Res. 2019 Feb;109:76-88. doi: 10.1016/j.jpsychires.2018.11.017. Epub 2018 Nov 22. PMID 30508746
- [Result] Levis B, Benedetti A, Thombs BD; DEPRESsion Screening Data (DEPRESSD) Collaboration. Accuracy of Patient Health Questionnaire-9 (PHQ-9) for screening to detect major depression: individual participant data meta-analysis. BMJ. 2019 Apr 9;365:l1476. doi: 10.1136/bmj.l1476. PMID 30967483
- [Result] Swenson JR. Quality of life in patients with coronary artery disease and the impact of depression. Curr Psychiatry Rep. 2004 Dec;6(6):438-45. doi: 10.1007/s11920-004-0008-x. PMID 15538992
- [Result] Rudisch B, Nemeroff CB. Epidemiology of comorbid coronary artery disease and depression. Biol Psychiatry. 2003 Aug 1;54(3):227-40. doi: 10.1016/s0006-3223(03)00587-0. PMID 12893099